CLINICAL TRIAL: NCT05825196
Title: Study of Serum Tumor Markers of HBV Associated HCC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YXLL-KY-2023(026)
Record Dates: First submitted 2023-03-26; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: HCC
Keywords: HBV related HCC
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Paired tumor, adjacent non-tumor liver tissues and blood samples from a cohort of HBV-related HCC patients, and blood samples from healthy subjects were selected as control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HBV-associated HCC group: The patient was finally diagnosed with HBV-related HCC by examination and imaging examination, and the clinicopathologic data were complete.
  Interventions: Diagnostic Test: tumor tissue and blood tests
- negative control group: HBV positive but not HCC
  Interventions: Diagnostic Test: tumor tissue and blood tests
- Healthy control group: Healthy crowd
  Interventions: Diagnostic Test: tumor tissue and blood tests

INTERVENTIONS:
Diagnostic Test: tumor tissue and blood tests — In this study, we need to collect an extra tube of blood for routine testing and the tissue after completion of pathological examination.

SUMMARY:
In this study, the investigators will detect the expression of four potential HBV-related HCC biomarkers: PGIR,FAM3C,LAMB1 and SDC4 in tumor tissues and peripheral blood, to explore the specific molecular markers for the early diagnosis of HBV-related HCC.

DETAILED DESCRIPTION:
Paired hepatitis B virus (HBV)-related hepatocellular carcinoma (HCC) and adjacent liver tissues were selected, and the mRNA and protein expressions of the PGIR,FAM3C,LAMB1 and SDC4 biomarkers in tissues were detected by RT-PCR, western Blot and immunohistochemical analysis. At the same time, healthy subjects were selected as the control group, and mRNA and protein expression levels of the above molecules in blood were detected by RT-PCR and ELISA. At the same time, the correlation between the above biomarkers and the clinical data of patients, such as diagnosis, pathological grading, recurrence, metastasis and survival time was statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* No local or systemic treatment was performed before surgery. The patients were finally diagnosed with HBV-related HCC by examination and imaging examination, and the clinicopathologic data were complete.

Exclusion Criteria:

* Patients with benign liver diseases, such as hepatic cysts and hepatic hemangiomas, or have tumors other than HBV-related HCC.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the patients admitted to the First Affiliated Hospital of Shandong First Medical University
Sampling Method: Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of RNA and protein for diagnosis | 6 months
  Detect the content of the RNA and protein in tumor and serum

IPD SHARING:
Plan to Share IPD: No